CLINICAL TRIAL: NCT03619421
Title: Evaluation of Zinc Supplementation Taken Prior or With Food
Brief Title: Zinc Supplement Before or With Food in Generally Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CHO23
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2018-08

CONDITIONS: Zinc Deficiency; Dyslipidemias; Zinc Excess; Inflammation
Keywords: zinc; nutrition; supplement; food
MeSH Terms: conditions — Dyslipidemias; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Random number used to label samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement with food (Experimental): Zinc supplement to be taken at time of breakfast consumption
  Interventions: Dietary Supplement: Zinc supplement
- supplement prior to food (Experimental): Zinc supplement to be taken 30-min before breakfast consumption
  Interventions: Dietary Supplement: Zinc supplement

INTERVENTIONS:
Dietary Supplement: Zinc supplement — 25 mg

SUMMARY:
The purpose of this study is to determine the influence of food consumption timing on the body's response to a zinc supplement

DETAILED DESCRIPTION:
This research is a dietary intervention study designed to evaluate the effect of the food consumption timing on the absorption of zinc supplement.

The main objective is to measure plasma zinc in generally healthy male subjects, who will consume zinc supplement with food or 30-min before food for 2-weeks.

In addition to the primary objectives, correlations in enzyme activity with changes in fat metabolism, namely circulating triglyceride and cholesterol, will be determined. This will enable the determination of the effect of a low Zn intake on various aspects of dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* willing to stop supplementation 4 weeks prior to start of the study
* has an operative understanding of English
* no plans to move from the area during the study period
* regularly eat breakfast

Exclusion Criteria:

* Chronic or acute metabolic disease
* smoker or user of nicotine products
* history of alcohol abuse, or use of illicit drugs (incl marijuana)
* Is underweight or overweight, body mass index (BMI) < 18 or > 30 kg/m2

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Plasma Zinc changes | Day 0, Day 15
  Change in plasma zinc

SECONDARY OUTCOMES:
Body weight changes | Day 0, Day 15
  Body weight changes
Essential Fatty acid changes | Day 0, Day 15
  Essential Fatty acid changes
Blood glucose changes | Day 0, Day 15
  Blood glucose changes

CONTACTS AND LOCATIONS:
Overall Officials: Jung Suh, PhD, Principal Investigator — UCSF Benioff Children's Hospital Oakland Research Institute
Locations (1):
- UCSF Benioff Children's Hospital Oakland Research Institute, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massih YN, Hall AG, Suh J, King JC. Zinc Supplements Taken with Food Increase Essential Fatty Acid Desaturation Indices in Adult Men Compared with Zinc Taken in the Fasted State. J Nutr. 2021 Sep 4;151(9):2583-2589. doi: 10.1093/jn/nxab149. PMID 34236435